CLINICAL TRIAL: NCT03408405
Title: ADRENL - ACTHAR Gel for Drug REsistant Nephrotic Syndrome in Children, Pilot Study
Brief Title: ACTHAR Gel for Drug REsistant Nephrotic Syndrome in Children
Acronym: ADRENL
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Withdrawal of funding from primary sponsor
Sponsor: Rhode Island Hospital (Other)
Collaborators: Mallinckrodt (Industry); University of Minnesota (Other); Medalytics (Unknown)
Responsible Party: Principal Investigator, Mohammed Khurram Faizan, Principal Investigator, Rhode Island Hospital
Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 1050945-5
Record Dates: First submitted 2018-01-08; First posted 2018-01-24 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Steroid-Resistant Nephrotic Syndrome
MeSH Terms: conditions — Nephrotic Syndrome

STUDY DESIGN:
Intervention Model Description: Inclusion Criteria:
  1. Patients between the ages of 2-21 years who fail a minimum of 12 weeks of cumulative therapy with prednisone OR one other alternate immunosuppressive agent for treatment of nephrotic syndrome, will be eligible for inclusion. Nephrotic syndrome is defined as: Presence of edema, Edema, UP/C ≥2, ≥300mg/dl or 3+ protein on Albustix, and hypoalbuminemia ≤2.5 g/dL
  2. Calculated GFR (eGFR) using modified Schwartz formula of > 50 mls/min/m2. (Modified Schwartz formula = 0.413 x height (cms) ÷ serum creatinine mg/dL)
  3. A clinical or biopsy diagnosis of nephrotic syndrome within the last 3 years prior to enrollment in the study.
  4. Renal biopsy (if available) consistent with a diagnosis of Minimal Change Disease, IgM nephropathy, Mesangioproliferative Glomerulonephritis, Primary Focal Segmental Glomerulosclerosis or C1q Nephropathy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Acthar Gel treatment group (Experimental): Participants will be treated with 'Acthar Gel 80 UNT/ML Injectable Solution'. Initial dose for week 1 will be 50% of 80 units, injected twice per week. Week 2 is 75% of 80 units, week 3 and throughout treatment period (6 months in total) will be 80 units/ml twice per week.
  Interventions: Drug: Acthar Gel 80 UNT/ML Injectable Solution

INTERVENTIONS:
Drug: Acthar Gel 80 UNT/ML Injectable Solution — Participant will self inject 'Acthar Gel 80 UNT/ML Injectable Solution' 2 x per week for six months.
  Other Names: H.P. Acthar gel

SUMMARY:
We propose to study the use of purified porcine Acthar Gel (ACTHAR, Mallinckrodt Pharmaceuticals) for treatment of steroid resistance nephrotic syndrome (SRNS) in a prospective pilot study. We plan to enroll 25 children between the ages of 2 to 21 years. Children fulfilling strict inclusion criteria, whose parents agree to written informed consent after institutional IRB approval for the study, will be enrolled. Purified porcine Acthar Gel will be administered SQ to all children using a defined treatment protocol for a period of six months. Renal function, urine protein excretion, serum albumin levels, blood pressure and growth parameters will be monitored closely on all patients. Baseline urine protein excretion will be compared to end of treatment levels to determine successful response to therapy. There will be an 18 month enrollment period, 6 month treatment period and a 12 month follow-up period.

DETAILED DESCRIPTION:
Treatment Protocol:

Patients who fulfill inclusion criteria and who agree to participate after signing informed consent and assent forms will be treated with the following protocol:

Acthar Gel will be dosed by body surface area (BSA) using the Dubois Method. The dose of Acthar Gel will be 80 units/1.73 m2 per dose administered subcutaneously (SQ) twice a week on Mondays and Thursdays.

Week 1 to 2:

During week 1, patients will receive 50% of initial calculated dose twice a week.

During week 2, patients will receive 75% of initial calculated dose twice a week.

Week 3 to 6 Months:

Patients will receive the full dose of Acthar Gel (80 units/1.73 m2 per dose) administered subcutaneously (SQ) twice a week on Mondays and Thursdays.

During this period, the treating physician will have the discretion of reducing the dose of Acthar Gel by 25-50% based on response with respect to reduction in proteinuria and tolerability of side-effects (uncontrolled hypertension, excessive weight gain, severe acne, hyperglycemia, etc.)

Patients will have the option of remaining on Acthar Gel after the 6 month study period based on clinical response at discretion of the co-PI. Study drug will be provided free of cost to patients in the first 6 months only.

Concomitant Treatments:

1. Amlodipine 0.1 mg/kg PO in one or two divided doses will be given to all patients who develop elevated blood pressure (>95th percentile) starting after 14 days of initiation of Acthar Gel therapy and will continue till 6 months. Dose can be increased up to 0.5 mg/kg divided bid as needed to achieve goal BP <95th percentile. If Amlodipine is not covered by the participants insurance, then an alternate calcium channel blocker will be started at the clinical discretion of the PI/co-PI that is covered by insurance. If the participant is not covered by any insurance the participant will have to pay out of pocket
2. If BP remains elevated despite maximum calcium channel therapy as described in the study protocol above, the choice and dose of additional anti-hypertensive agents will be at the discretion of the study investigator on an individualized and as needed basis.
3. Patients on prednisone on initiation of study will be tapered off over 2-4 weeks. Non-steroidal immunosuppression may be tapered off over four weeks after the start of Acthar Gel therapy at the discretion of the PI/Co-PI.
4. Additional standard of care therapy (statins, vitamin D, antacids, etc.) can be continued and modified based on the discretion and clinical judgment of the study PI/Co-PIs.

Quality of Life Assessment:

Quality of life will be measured using the patient and parent self-report versions of the Pediatric Quality of Life Inventory, ESRD, Acute Version. The PedsQL 3.0 ESRD Scales measure physical, emotional, social and role (i.e. school) dimensions. Scores are derived for physical functioning and psychological functioning, in addition to a total score, which enables comparison against healthy populations. Scales are rated on a 5-point Likert scale (0 = never, 1= almost never, 2 = sometimes, 3 = often, 4 = almost always), with scores linearly transformed to range from 0 - 100, with higher scores indicating fewer problems or symptoms.

Surveys will be administered by trained study personnel at enrollment (baseline), six months, 12 months, and 18 months.

Laboratory Testing:

Baseline and then once a month till the end of the treatment period (6 months): Serum electrolytes, BUN, creatinine, albumin, ACTH level, glucose, random cortisol, calcium, magnesium, phosphorus, ALT, AST, total and direct bilirubin, fasting cholesterol, triglycerides, HDL, LDL, urine protein to creatinine ratio. During the 12 month follow-up period laboratory evaluation will be performed every third month. (11 total blood draws). A urine pregnancy test shall be sent on all female patients of child-bearing potential at the beginning and end of treatment period.

All available biopsy slides will be reviewed by a blinded renal pathologist to insure accuracy and to confirm the initial histologic diagnosis.

Telephone Contact One, two and three weeks after initial dose. Phone contacts will screen for: adverse events, and review dosing of ACTHAR GEL.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between the ages of 2-21 years who fail a minimum of 12 weeks of cumulative therapy with prednisone OR one other alternate immunosuppressive agent for treatment of nephrotic syndrome, will be eligible for inclusion. Nephrotic syndrome is defined as: Presence of edema, Edema, UP/C ≥2, ≥300mg/dl or 3+ protein on Albustix, and hypoalbuminemia ≤2.5 g/dL
2. Calculated GFR (eGFR) using modified Schwartz formula of > 50 mls/min/m2. (Modified Schwartz formula = 0.413 x height (cms) ÷ serum creatinine mg/dL)
3. A clinical or biopsy diagnosis of nephrotic syndrome within the last 3 years prior to enrollment in the study.
4. Renal biopsy (if available) consistent with a diagnosis of Minimal Change Disease, IgM nephropathy, Mesangioproliferative Glomerulonephritis, Primary Focal Segmental Glomerulosclerosis or C1q Nephropathy

Exclusion Criteria:

1. Patients with an inherited or genetic disorder presenting with nephrotic syndrome (eg: NPHS 1 & 2 defects, WT-1 mutations, α actinin 4 mutation, TRP-6 mutation).
2. Presence of diabetes or severe (stage 2) uncontrolled hypertension.
3. Any metabolic condition that specifically precludes the use of Acthar Gel for treatment.
4. Pregnancy or unwilling to agree to contraception which may include abstinence.
5. eGFR <50 mls/min/m2

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Remission of proteinuria | 18 months
  Partial remission: Greater than or equal to 50% reduction in proteinuria when compared to baseline.
  Complete remission: Greater than or equal to 90% reduction in proteinuria when compared to baseline or Urine Protein Creatinine ratio less than 0.5.

SECONDARY OUTCOMES:
Blood pressure | 18 months
  Blood pressure during study visit as measured in mm/Hg
Serum Creatinine | 18 months
  Serum value in mg/dL
BMI | 18 months
  Weight (kgs) and height (cms) will be combined to report BMI in kg/m^2
Serum Glucose | 18 months
  Serum value in mg/dL
Serum Lipids | 18 months
  Serum Value in mg/dL
Quality of life measures obtained via survey | 18 months
  PedsQL 3.0 will be used as the standardized survey tool

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed K Faizan, MD, Principal Investigator — Rhode Island Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coppo R. Non-steroidal and non-cytotoxic therapies for nephrotic syndrome. Nephrol Dial Transplant. 2008 Jun;23(6):1793-6. doi: 10.1093/ndt/gfn211. Epub 2008 Apr 25. No abstract available. PMID 18441003
- [Background] Mackay MT, Weiss SK, Adams-Webber T, Ashwal S, Stephens D, Ballaban-Gill K, Baram TZ, Duchowny M, Hirtz D, Pellock JM, Shields WD, Shinnar S, Wyllie E, Snead OC 3rd; American Academy of Neurology; Child Neurology Society. Practice parameter: medical treatment of infantile spasms: report of the American Academy of Neurology and the Child Neurology Society. Neurology. 2004 May 25;62(10):1668-81. doi: 10.1212/01.wnl.0000127773.72699.c8. PMID 15159460
- [Background] Rauen T, Michaelis A, Floege J, Mertens PR. Case series of idiopathic membranous nephropathy with long-term beneficial effects of ACTH peptide 1-24. Clin Nephrol. 2009 Jun;71(6):637-42. doi: 10.5414/cnp71637. PMID 19473632
- [Background] Ponticelli C, Passerini P, Salvadori M, Manno C, Viola BF, Pasquali S, Mandolfo S, Messa P. A randomized pilot trial comparing methylprednisolone plus a cytotoxic agent versus synthetic adrenocorticotropic hormone in idiopathic membranous nephropathy. Am J Kidney Dis. 2006 Feb;47(2):233-40. doi: 10.1053/j.ajkd.2005.10.016. PMID 16431252
- [Background] Berg AL, Arnadottir M. ACTH-induced improvement in the nephrotic syndrome in patients with a variety of diagnoses. Nephrol Dial Transplant. 2004 May;19(5):1305-7. doi: 10.1093/ndt/gfh110. No abstract available. PMID 15102969
- [Background] Bomback AS, Tumlin JA, Baranski J, Bourdeau JE, Besarab A, Appel AS, Radhakrishnan J, Appel GB. Treatment of nephrotic syndrome with adrenocorticotropic hormone (ACTH) gel. Drug Des Devel Ther. 2011 Mar 14;5:147-53. doi: 10.2147/DDDT.S17521. PMID 21448451
- [Background] Bomback AS, Canetta PA, Beck LH Jr, Ayalon R, Radhakrishnan J, Appel GB. Treatment of resistant glomerular diseases with adrenocorticotropic hormone gel: a prospective trial. Am J Nephrol. 2012;36(1):58-67. doi: 10.1159/000339287. Epub 2012 Jun 19. PMID 22722778
- [Background] LAUSON HD, FORMAN CW, McNAMARA H, MATTAR G, BARNETT HL. The effect of corticotropin (ACTH) on glomerular permeability to albumin in children with the nephrotic syndrome. J Clin Invest. 1954 Apr;33(4):657-64. doi: 10.1172/JCI102936. No abstract available. PMID 13152205